CLINICAL TRIAL: NCT03803319
Title: Microbiological and Physiological Effects of Dietary Supplementation With Fibre in Irritable Bowel Syndrome: a Randomised Controlled Trial
Brief Title: Effects of Dietary Fibre in Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Universidad Veracruzana (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18/WA/0313
Record Dates: First submitted 2018-12-14; First posted 2019-01-14 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: dietary fibre
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: multi-centre, 3 treatment, placebo-controlled trial
Who Masked: Participant, Investigator
Masking Description: Participants and Investigators will be blinded to the fibre provided over the 8-week intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fibre 1 (combined fibres) (Active Comparator): Ingestion of 150mls water with 7.5g fibre (two times a day)
  Interventions: Dietary Supplement: Fibre 1 (combined fibres)
- Fibre 2 (natural fibres) (Active Comparator): Ingestion of 150mls water with 15g fibre (two times a day)
  Interventions: Dietary Supplement: Fibre 2 (natural fibres)
- Dietary Supplement (placebo) (Placebo Comparator): Ingestion of 150mls water with 7.5g (two times a day)
  Interventions: Dietary Supplement: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Fibre 1 (combined fibres) — Dietary fibre supplement
  Arms: Fibre 1 (combined fibres)
Dietary Supplement: Fibre 2 (natural fibres) — Dietary fibre supplement
  Arms: Fibre 2 (natural fibres)
Dietary Supplement: Dietary Supplement: placebo — Dietary supplement
  Arms: Dietary Supplement (placebo)

SUMMARY:
The aim of the study is to investigate how different dietary fibre combinations affects physiological and microbiological outcomes, in addition to symptoms in those with IBS. The study will also explore the differences in responses between different fibres in different sub-types of IBS (e.g. constipation-predominant, diarrhoea-predominant and mixed).

DETAILED DESCRIPTION:
Currently, national and international guidelines are based upon trials of dietary fibre in IBS symptoms that report opposing effects. For this reason, recommendations regarding dietary fibre food supplementation in IBS are often conflicting. Indeed, the confusion surrounding dietary fibre recommendations in IBS is a consequence of the limited understanding of the different types of dietary fibres used, their physiology and their functions in different sub-groups of IBS.

Different fibres have different characteristics (e.g. solubility, viscosity and fermentability) which drive different functionalities (stool forming, fermentation) in the gastrointestinal tract, yet it is currently unknown whether administration of dietary fibre combinations will result in symptomatic improvement in people with IBS.

Participants will be randomised to one of three parallel arms for a duration of 8 weeks.

The study will consist of 4 visits in total. The first visit will involve taking consent and assessing eligibility. Participants will complete the Rome IV diagnostic criteria as part of their eligibility assessment. Participants will be asked to complete a food and symptom diary for the next 7 days. Diary data will be used to confirm frequency and severity of IBS symptoms and ensure there is no discrepancy between participant report on the Rome IV diagnostic criteria.

Visit 2: Baseline (approx 1.5 hours). Height and weight will be recorded. Participants will complete 7 questionnaires, provide a stool sample, a blood sample and will ingest the SmartPill (wireless motility capsule). Participants will blinded to the intervention and will be provided with sachets containing either fibre 1 (combined fibres), fibre 2 (natural fibres) or placebo to consume over an 8-week period.

Visit 3: Mid-point (approx 1 hour). Participants will complete 5 questionnaires and provide a stool sample.

Visit 4: Endpoint (approx 1.5 hours). Height and weight will be recorded. Participants will complete 7 questionnaires, provide a stool sample, a blood sample and will ingest the SmartPill (wireless motility capsule).

ELIGIBILITY:
Inclusion Criteria:

* Interested in taking part
* Ability to give informed consent
* Men and women aged 18-65 years with diarrhoea-predominant IBS (IBS-D), constipation-dominant IBS (IBS-C), or mixed (IBS-M), based on fulfilment of the Rome IV criteria for irritable bowel syndrome who do not have a major medical condition (e.g. diabetes, psychiatric or current eating disorders), severe oesophagitis, gastritis or duodenitis, gastrointestinal disease (inflammatory bowel disease, coeliac disease, active diverticulitis), or history of previous GI surgery (excluding appendicectomy, cholecystectomy and haemorrhoidectomy), severe renal, cardiac, pulmonary, or other chronic diseases likely to affect motility, history of gastric bezoars.

Exclusion Criteria:

* Females who report to be pregnant or lactating
* Body Mass Index (BMI) >40 kg/m2
* Use of unpermitted medications in the last 4 weeks prior to, or during the study including: Antibiotics within the last 4weeks, dietary fibre food supplements within the last 4 weeks (e.g. Fybogel, Lactulose), prebiotics or probiotics (in food products or as supplements) within the last 4 weeks, other dietary supplements that may affect the luminal microenvironment of the intestine (e.g. Orlistat)
* Use of drugs known to alter GI motility, transit or gastric pH (e.g. mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines) in the last 1 week
* Full bowel preparation for a diagnostic procedure within the last 4 weeks
* Changes to IBS medications or dose in the 4 weeks prior to the study
* Changes to anti-depressant medications or dose in the 12 weeks prior to the study
* Swallowing disorders (physical or psychological)
* Use of implantable and/or medical devices such as pacemakers
* Individuals following extreme diets e.g. 8 or more caffeinated serves per day, 4 or more bottles of wine (40 or more units of alcohol per week) or equivalent per week as assessed by diet questionnaires or changes to smoking habits
* Individuals who have participated in other intervention trials within 3 months prior to screening
* Allergies to components (soy) of the SmartBar (required for SmartPill protocol)
* Abdominal pain for less than 2 days in the screening week (based on the GSRS mild to severe)
* Those who report adequate relief of symptoms at baseline using the GSQ

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-01-11 (Actual); Study Completion 2020-01-11 (Actual)

PRIMARY OUTCOMES:
Relative abundance of faecal bifidobacteria as assessed using 16S rRNA community profiling (Illumina Miseq) of bacterial genomic DNA isolated from stool samples | 0, 4, 8 weeks
  Change from baseline in relative abundance of bifidobacteria between the three groups at 8 weeks
IBS symptoms as assessed using the Global Symptom Question (GSQ) | 0, 4, 8 weeks
  Change from baseline in the GSQ between the three groups at 8 weeks

SECONDARY OUTCOMES:
Whole gut and regional gut transit time as assessed using a telemetric device (wireless motility capsule: SmartPill) | 0 and 8 weeks
  Change from baseline in whole and regional gut transit time between the three groups at 8 weeks
Colonic pH units as assessed using a telemetric device (wireless motility capsule: SmartPill) | 0 and 8 weeks
  Change from baseline in colonic pH units between the three groups at 8 weeks
Pressure (mmHg) as assessed using a telemetric device (wireless motility capsule: SmartPill) | 0 and 8 weeks
  Change from baseline in pressure (mmHg) between the three groups at 8 weeks
Faecal short-chain fatty acids (SCFAs) as assessed using gas-liquid chromatography | 0, 4, 8 weeks
  Change from baseline in microbial metabolites between the three groups at 8 weeks
Faecal gut microbiota (α and β diversity) as assessed using 16S rRNA community profiling (Illumina Miseq) of bacterial genomic DNA isolated from stool samples | 0, 4, 8 weeks
  Change from baseline in faecal gut microbiota (α and β diversity) between the three groups at 8 weeks
Faecal volatile organic compounds (VOCs) as assessed using gas chromatography sensor device | 0 and 8 weeks
  Change from baseline in VOCs between the three groups at 8 weeks
Serum/plasma appetite hormones (ghrelin, pg/ml) as determined by enzyme-linked immunosorbent assay (ELISA) | 0 and 8 weeks
  Change from baseline in ghrelin concentrations between the three groups at 8 weeks
Serum/plasma (leptin, pg/ml) as determined by enzyme-linked immunosorbent assay (ELISA) | 0 and 8 weeks
  Change from baseline in leptin concentrations between the three groups at 8 weeks
Serum/plasma metabolites as determined using metabolomics | 0 and 8 weeks
  Change from baseline in plasma/serum metabolites between the three groups at 8 weeks
Stool consistency as assessed using the Bristol Stool Form Scale (BSFS) (7 point scale; Type 1 to Type 7) | 0 and 8 weeks
  Change from baseline in stool consistency and stool frequency between the three groups at 8 weeks
Gastrointestinal symptoms as assessed using the Gastrointestinal Symptom Rating Scale (GSRS) over 7 days (absent - severe) | 0 and 8 weeks
  Change from baseline in gastrointestinal symptoms between the three groups at 8 weeks
Gastrointestinal symptoms as assessed using the Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS) (visual analogue scale: no pain - severe) | 0, 4, 8 weeks
  Change from baseline in the severity of gastrointestinal symptoms between the three groups at 8 weeks
Quality of Life (QoL) general as assessed using the SF-36 | 0, 4, 8 weeks
  Change from baseline in general QoL between the three groups at 8 weeks
Disease-specific QoL as assessed using the IBS-QoL (5 point scale: not at all - a great deal) | 0, 4, 8 weeks
  Change from baseline in disease-specific QoL between the three groups at 8 weeks
Perceived stress as assessed using the Perceived Stress Score (PSS) (5 point scale: never- very often) | 0, 4, 8 weeks
  Change from baseline in perceived stress between the three groups at 8 weeks
Dietary fibre acceptability as assessed using an acceptability questionnaire (5 point scale: not at all acceptable - extremely acceptable) | 8 weeks
  Dietary fibre acceptability between the three groups at 8 weeks
Nutrient intake as assessed using a 7-day food diary | 0 and 8 weeks
  7-day food diary
Physical activity as assessed using the International Physical Activity Questionnaire (IPAQ) | 0 weeks
  Physical activity
Waist circumference as assessed using a standard measuring tape (inches) | 0 and 8 weeks
  Change from baseline in waist circumference between the three groups at 8 weeks
Hydrogen/methane breath testing as assessed using the Gastrocheck Gastrolyzer V9.0 in parts per million | 0 and 8 weeks
  Hydrogen/methane breath testing

OTHER OUTCOMES:
Visceral sensitivity as assessed using the Visceral Sensitivity Index (VSI) (6 point scale: strongly agree - strongly disagree) | 0 and 8 weeks
  Change from baseline in visceral sensitivity between the three groups at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Whelan, PhD, Study Director — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participant information will only be available to the Investigators undertaking the study.